CLINICAL TRIAL: NCT03152006
Title: Adolescent Coordinated Transition (ACT) to Improve Health Outcomes Among Nigerian HIV+ Youth
Brief Title: Adolescent Coordinated Transition Nigerian HIV+ Youth
Acronym: ACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Echezona Ezeanolue, Professor of Public Health and Pediatrics, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 990070-4; R01HD089871 (NIH)
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: HIV/AIDS
Keywords: Healthcare transition; Adolescents; Nigeria
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control arm does not receive the ACT intervention.
- ACT Intervention (Experimental): Intervention activities include the three components of the ACT intervention: (1) alternating pediatric and adult clinic visits in the 12 month pre-transfer period (2) peer facilitated organized support group during the 24-month graduated transition period and (3) patient advocate and case management team to coordinate transfer process.
  Interventions: Other: ACT

INTERVENTIONS:
Other: ACT — Coordinated, graduated transition which includes an early introduction to the adult clinician during the PAPA pre-transfer period, a peer-facilitated organized support group aimed at improving transition readiness and addressing critical psychosocial skills including self-efficacy and locus of control and a case management team including a patient advocate who coordinates the transfer between pediatric and adult care teams.
  Arms: ACT Intervention

SUMMARY:
The purpose of this study is to evaluate the comparative effectiveness of a comprehensive, coordinated transition protocol which includes an early introduction to the adult provider, an integrated case management team and a peer-facilitated organized support group on retention in care, viral suppression and psychosocial wellbeing among adolescents living with HIV.

DETAILED DESCRIPTION:
Using a two-arm cluster randomized design, our proposed study will evaluate the comparative effectiveness of ACT, a coordinated protocol for transitioning adolescents living with HIV (ALHIV) from pediatric to adult care (Intervention Group; IG) versus the usual abrupt transfer to adult care (Control group; CG) on rates of retention in care and viral suppression, and differences in perceived psychosocial wellbeing. Twelve health facilities, two in each of the six geopolitical zones of Nigeria will be pair-matched and randomly assigned to either IG (N=6 health facilities) or CG (N=6 health facilities). A total of 216 ALHIV will be enrolled in the study over a 36-month period. The primary outcome will be the difference in the rate of retention between the groups. Secondary outcomes will be difference in the rate of viral suppression and the difference in perceived psychosocial wellbeing. Additionally, the investigators will conduct mediation/moderation analysis to examine the role of intermediate variables such as transition readiness, perceived mental health, social support, health locus of control, self-esteem and sexual risk behavior self-efficacy on the primary outcomes. Implementation factors will be assessed using the hybrid 2 model.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* Aware of HIV diagnosis
* Currently on ART

Exclusion Criteria:

* Medically unstable

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 216 (Estimated)
Dates: Start 2017-06-28 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Retention in care in care 6 months post-transfer | 6 months
  Proportion of participants who had at least 1 clinical visit to an HIV provider within the 6 months post-transfer
Retention in care 12 months post-transfer | 12 months
  Proportion of participants who had at least 2 clinical visits to an HIV provider separated by 6 months within the 1 year period post-transfer
Retention in care 24 months post-transfer | 24 months
  Proportion of participants who had at least 2 clinical visits to an HIV provider separated by 6 months within a 1 year period during the second year post-transfer

SECONDARY OUTCOMES:
Viral Suppression | Enrollment, baseline (12 months), 24 and 36 months
  Proportion of participants with undetectable viral load
Mental Health and Wellbeing | Enrollment, baseline (12 months), 24 and 36 months
  Mental health continuum-short form Questionnaire
Health Locus of Control | Enrollment, baseline (12 months), 24 and 36 months
  Health Locus of control / Self-esteem Questionnaire
Social Support | Enrollment, baseline (12 months), 24 and 36 months
  Functional Social Support Questionnaire
Sexual Risk Behavior | Enrollment, baseline (12 months), 24 and 36 months
  Sexual Risk Beliefs and Behavior Self Efficacy Questionnaire
Transition Readiness | Enrollment, baseline (12 months), 24 and 36 months
  Transition Readiness Assessment Questionnaire

CONTACTS AND LOCATIONS:
Locations (5):
- Nigeria (5):
  - Institute of Human Virology, Abuja, Federal Capital Territory
  - Center for Integrated Health Program, Abuja
  - Centre for Clinical Care and Research, Abuja
  - Family Health International, Abuja
  - AIDS Prevention Initiative Nigeria, Lagos

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sam-Agudu NA, Pharr JR, Bruno T, Cross CL, Cornelius LJ, Okonkwo P, Oyeledun B, Khamofu H, Olutola A, Erekaha S, Menson WNA, Ezeanolue EE. Adolescent Coordinated Transition (ACT) to improve health outcomes among young people living with HIV in Nigeria: study protocol for a randomized controlled trial. Trials. 2017 Dec 14;18(1):595. doi: 10.1186/s13063-017-2347-z. PMID 29237487